CLINICAL TRIAL: NCT07220421
Title: Evaluate Foundational Wellness Programs to Help Reduce Clinician Burnout and Improve Professional Fulfilment in Health Care Professionals.
Brief Title: Foundational Programs to Combat Clinician Stress
Acronym: FACCTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 857510
Record Dates: First submitted 2025-09-02; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Burnout, Professional; Stress, Psychological; Stress, Physiological; Psychological Well-Being; Mind-Body Therapies; Work Related Stress
Keywords: Sudarshan Kriya Yoga (SKY) Breathing and Sahaj Meditation; Stress Reduction; Healthcare Professional Burnout; Workplace Wellbeing; Work Life Balance; Physician; Healthcare Provider; Cognitive Performance; Cognitive Attention; Depression; Anxiety; Sleep; Heart Rate Variability; Resilience; Social Connection; Self-Valuation; Professional Fulfilment; Medical Errors; Physician Turnover; Healthcare Economics; Occupational Burnout
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological; Psychological Well-Being; Occupational Stress; Respiratory Aspiration; Depression; Anxiety Disorders | interventions — Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sudarshan Kriya Yoga (SKY) Breathing and Sahaj Meditation (Experimental): The SKY Breathing and Sahaj Meditation program involves teaching cyclical breathing techniques with various hand positions and a Guided Meditation practice. This program also includes teaching Cognitive Reframing Tools (CRTs) for emotional regulation.
  Interventions: Behavioral: Sudarshan Kriya Yoga (SKY) Breathing and Sahaj Meditation
- Health Education Program (HEP) (Active Comparator): The Health Education Program (HEP) curriculum reviews various health related topics and facilitates group discussion on such topics. This program includes teachings on topics such as mental health, exercise and nature, nutrition and hydration, and self-care. It provides a learning experience on health topics and gives participants skills, tools, and knowledge to live healthier lives.
  Interventions: Other: Health Education Program (HEP)

INTERVENTIONS:
Behavioral: Sudarshan Kriya Yoga (SKY) Breathing and Sahaj Meditation — The SKY intervention is comprised of a week of baseline HRV and sleep metric readings, followed by an onboarding week of 3-day, 3.5 hours/day, online SKY workshops with a live instructor (10.5 hours total), followed by weekly online follow-up sessions with a live instructor (1 hour each) for a period of 4 weeks. Clinicians also practice on their own daily for 45 minutes during these 4 weeks and wear an Oura Ring continuously. They do not have to do their daily practice on the days that they have a follow-up session.
  Well-being and burnout metrics will be assessed using PFI Week 1, Week 4, and Week 6. Evaluation of the impact of the program on other factors as measured by other questionnaires Week 1 and Week 6. HRV and sleep metrics will be used as a physiologic marker of well-being and will be measured continuously via Oura Ring.
  Arms: Sudarshan Kriya Yoga (SKY) Breathing and Sahaj Meditation
Other: Health Education Program (HEP) — The HEP coaches will provide these sessions online with an initial onboarding week of 2-day, 3 hours/day online HEP workshop followed by weekly online follow up sessions for 2 hours each with a live instructor. They will also pursue 45 min of daily practice for a period of 4 weeks. They do not have to do their daily practice on the days that they have a follow-up session.
  Well-being and burnout metrics will be assessed using PFI Week 1, Week 4, and Week 6. Evaluation of the impact of the program on other factors as measured by other questionnaires Week 1 and Week 6. HRV and sleep metrics will be used as a physiologic marker of well-being and will be measured continuously via Oura Ring.
  Arms: Health Education Program (HEP)

SUMMARY:
This is a prospective, randomized, controlled clinical trial in which clinicians from University of Pennsylvania Health Systems (UPHS) including Penn Medicine- Lancaster General Health (LGH) and Massachusetts General Hospital (MGH) are offered a well-known program to help reduce clinician burnout: Sudarshan Kriya Yoga (SKY) Breathing and Sahaj Meditation Intervention.

DETAILED DESCRIPTION:
This study will not only measure psychometric data and cognitive metrics for clinician burnout but also assess physiological marker of wellbeing by collecting Heart Rate Variability (HRV) data and sleep scores. We expect to see significant improvement in psychophysiologic metrics including depression, anxiety, sleep problems, cognitive overload, mindfulness and heart rate variability.

The proposed prospective, randomized clinical trial will examine the effects of SKY in a large group of health care clinicians (physician, Advanced Practice Provider (APP), Certified Registered Nurse Practitioner (CRNP), Physician Assistant (PA), psychologist) within the US, examining the above constructs. Clinicians will be randomized one of 2 arms: SKY or an active control group.

This research initiative will enroll 90 clinicians in the SKY program. The SKY intervention is comprised of a week of baseline HRV and sleep metric readings, followed by an onboarding week of 3-day, 3.5 hours/day, online SKY workshops with a live instructor (10.5 hours total), followed by weekly online follow-up sessions with a live instructor (1 hour each) for a period of 4 weeks. Clinicians also practice on their own daily for 45 minutes during these 4 weeks and wear an Oura Ring continuously. They do not have to do their daily practice on the days that they have a follow-up session.

90 clinicians will be assigned as controls and participate in an active control group with Health Education Program (HEP). The HEP coaches will provide these sessions online with an initial onboarding week of 2-day, 3 hours/day online HEP workshop followed by weekly online follow up sessions for 2 hours each with a live instructor. They will also pursue 45 min of daily practice for a period of 4 weeks. They do not have to do their daily practice on the days that they have a follow-up session.

Well-being and burnout metrics will be assessed using Professional Fulfillment Index (PFI) collected at baseline (week 1), midpoint (week 4), and endpoint (week 6) in the SKY intervention and control group. HRV and sleep score will be used as physiologic markers of well-being and will be measured daily in the SKY and control groups. Secondary outcomes will be measured to evaluate the impact of the programs on other factors as measured by questionnaires at Week 1 and Week 6:

Depression (PROMIS 8a: 8-item Emotional Distress - Depression scale) Anxiety (PROMIS 8a: 8-item Emotional Distress - Anxiety scale) Sleep (PROMIS 8a: 8-item Sleep-Related Impairment scales) Intent to Leave (1 item) Self-Valuation (Stanford Self-Valuation Scale, 4 items) Stanford Impact of Work on Personal Relationships scale (IWPR, 4 items) Social Connectedness Scale-Revised (SCS-R; 20 items) Mindful Attention (5-item Mindful Attention Awareness Scale) Cognitive Errors (12-item Attention-Related Cognitive Errors Scale) Measurement of Self-Reported Medical Errors (SRME, 4 items)

The survey data will be statistically analyzed using linear mixed effects models. The goal of the project is to mitigate or reverse initial symptoms of clinician burnout with the SKY program at a statistically significant difference as compared to the control. The intended outcome is to implement the foundational wellness SKY program on a wider scale to other healthcare professionals

Further details about the study design and references can be found in the full study protocol, once uploaded.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 years of age,
* UPHS or MGH clinician (physician, APP, CRNP, PA, psychologist),
* Access to smart phone and internet,
* Ability to give informed consent,
* Interested in wearing an Oura ring and being part of a study to evaluate breath and meditation-derived exercises,
* Willing to do relaxation exercise every day for 4 weeks.

Exclusion Criteria:

* Currently maintaining a regular/daily mind-body program practice (eg. meditation, yoga or breathing techniques),
* Atrial fibrillation,
* Pacemaker/defibrillator,
* Untreated or severe obstructive sleep apnea (AHI>=30),
* History of diaphragm paralysis,
* Unable or unwilling to complete the workshop,
* Severe chronic obstructive pulmonary disease (COPD),
* Severe valvular heart disease,
* Prior or planned chest/abdominal or nasal/facial surgery within 6 months,
* Severe psychiatric illness (e.g. schizophrenia, schizoaffective disorder, bipolar disorder), active substance use, seizure disorder or major somatic illness (uncontrolled hypertension, lung disease, liver disease, cancer or heart disease).

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of well-being foundational programs on burnout in clinicians at hospital health systems utilizing the Stanford Professional Fulfilment Index. | Assess at Baseline (week1), Midpoint (week 4), and Endpoint (week 6).
  The unit of measurement for the Stanford Professional Fulfillment Index is Likert scale scores, reflecting how often the individual experiences aspects of fulfillment or burnout.
  These are ordinal scores with ranked responses, but the exact intervals between the scores are not numerically defined.

SECONDARY OUTCOMES:
Evaluation of Heart Rate Variability (HRV) as a physiologic metric for well-being in clinicians through continuous readings using the Oura Ring. | Daily for 6 weeks.
  Millisecond (ms) is the unit for HRV.
Evaluation of sleep scores as physiologic metrics for well-being in clinicians through continuous readings using the Oura Ring. | Daily for 6 weeks.
  Sleep score is a normalized score that ranges from 0 to 100, with 100 being the best possible score indicating ideal sleep quality.
Evaluation of the impact of the programs on depression as measure by the PROMIS 8a: 8-item Emotional Distress - Depression scale. | Assess at Baseline (week 1) and Endpoint (week 6).
  PROMIS 8a: 8-item Emotional Distress - Depression Scale: The score ranges from 8 to 40, and higher scores indicate worse depression.
Evaluation of the impact of the programs on anxiety as measure by the PROMIS 8a: 8-item Emotional Distress - Anxiety scale. | Assess at Baseline (week 1) and Endpoint (week 6).
  PROMIS 8a: 8-item Emotional Distress - Anxiety Scale: The score ranges from 8 to 40, and higher scores indicate worse anxiety.
Evaluation of the impact of the programs on sleep as measure by the PROMIS 8a: 8-item Sleep-Related Impairment scales. | Assess at Baseline (week 1) and Endpoint (week 6).
  PROMIS 8a: 8-item Sleep-Related Impairment Scale: The score ranges from 8 to 40, and higher scores indicate worse sleep-related impairment.
Evaluation of the impact of the programs on intent to leave place of employment as measure by the Intent to Leave 1 item scale. | Assess at Baseline (week 1) and Endpoint (week 6).
  Intent to Leave Scale (1 item): The score ranges from 1 to 5, and higher scores indicate stronger intent to leave.
Evaluation of the impact of the programs on self-valuation as measure by the Stanford Self-Valuation Scale, 4 items. | Assess at Baseline (week 1) and Endpoint (week 6).
  Stanford Self-Valuation Scale (4 items): The score ranges from 4 to 20, and higher scores indicate better self-esteem and self-worth.
Evaluation of the impact of the programs on impact of work on personal relationships as measure by the Stanford Impact of Work on Personal Relationships scale (IWPR, 4 items). | Assess at Baseline (week 1) and Endpoint (week 6).
  Stanford Impact of Work on Personal Relationships Scale (IWPR): The score ranges from 4 to 20, and higher scores indicate worse impact of work on personal relationships.
Evaluation of the impact of the programs on social connectedness as measure by the Social Connectedness Scale-Revised (SCS-R; 20 items). | Assess at Baseline (week 1) and Endpoint (week 6).
  Social Connectedness Scale-Revised (SCS-R; 20 items): The score ranges from 20 to 100, and higher scores indicate better social connectedness.
Evaluation of the impact of the programs on mindful attention as measure by the 5-item Mindful Attention Awareness Scale. | Assess at Baseline (week 1) and Endpoint (week 6).
  Mindful Attention Awareness Scale (MAAS, 5 items): The score ranges from 5 to 35, and higher scores indicate better mindfulness.
Evaluation of the impact of the programs on cognitive errors as measure by the 12-item Attention-Related Cognitive Errors Scale. | Assess at Baseline (week 1) and Endpoint (week 6).
  12-item Attention-Related Cognitive Errors Scale (ARCES): The score ranges from 12 to 60, and higher scores indicate more cognitive errors.
Evaluation of the impact of the programs on self-reported medical errors as measure by the Measurement of Self-Reported Medical Errors (SRME, 4 items). | Assess at Baseline (week 1) and Endpoint (week 6).
  Self-Reported Medical Errors Scale (SRME, 4 items): The score ranges from 4 to 20, and higher scores indicate more frequent medical errors.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Meesala, MD, Principal Investigator — Penn Medicine / Lancaster General Hospital
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Princeton Medical Center / Princeton Health affiliated sites, Plainsboro, New Jersey
  - Penn Medicine Lancaster General Health, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ligibel JA, Goularte N, Berliner JI, Bird SB, Brazeau CMLR, Rowe SG, Stewart MT, Trockel MT. Well-Being Parameters and Intention to Leave Current Institution Among Academic Physicians. JAMA Netw Open. 2023 Dec 1;6(12):e2347894. doi: 10.1001/jamanetworkopen.2023.47894. PMID 38100103
- [Background] Carriere JS, Cheyne JA, Smilek D. Everyday attention lapses and memory failures: the affective consequences of mindlessness. Conscious Cogn. 2008 Sep;17(3):835-47. doi: 10.1016/j.concog.2007.04.008. Epub 2007 Jun 15. PMID 17574866
- [Background] Osman A, Lamis DA, Bagge CL, Freedenthal S, Barnes SM. The Mindful Attention Awareness Scale: Further Examination of Dimensionality, Reliability, and Concurrent Validity Estimates. J Pers Assess. 2016;98(2):189-99. doi: 10.1080/00223891.2015.1095761. Epub 2015 Nov 11. PMID 26560259
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Trockel J, Bohman B, Wang H, Cooper W, Welle D, Shanafelt TD. Assessment of the Relationship Between an Adverse Impact of Work on Physicians' Personal Relationships and Unsolicited Patient Complaints. Mayo Clin Proc. 2022 Sep;97(9):1680-1691. doi: 10.1016/j.mayocp.2022.03.005. PMID 36058580
- [Background] Buysse DJ, Yu L, Moul DE, Germain A, Stover A, Dodds NE, Johnston KL, Shablesky-Cade MA, Pilkonis PA. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. Sleep. 2010 Jun;33(6):781-92. doi: 10.1093/sleep/33.6.781. PMID 20550019
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Trockel M, Bohman B, Lesure E, Hamidi MS, Welle D, Roberts L, Shanafelt T. A Brief Instrument to Assess Both Burnout and Professional Fulfillment in Physicians: Reliability and Validity, Including Correlation with Self-Reported Medical Errors, in a Sample of Resident and Practicing Physicians. Acad Psychiatry. 2018 Feb;42(1):11-24. doi: 10.1007/s40596-017-0849-3. Epub 2017 Dec 1. PMID 29196982
- [Background] Trockel M, Sinsky C, West CP, Dyrbye LN, Tutty M, Carlasare L, Wang H, Shanafelt T. Self-Valuation Challenges in the Culture and Practice of Medicine and Physician Well-being. Mayo Clin Proc. 2021 Aug;96(8):2123-2132. doi: 10.1016/j.mayocp.2020.12.032. Epub 2021 Jun 28. PMID 34210511
- [Background] Descilo T, Vedamurtachar A, Gerbarg PL, Nagaraja D, Gangadhar BN, Damodaran B, Adelson B, Braslow LH, Marcus S, Brown RP. Effects of a yoga breath intervention alone and in combination with an exposure therapy for post-traumatic stress disorder and depression in survivors of the 2004 South-East Asia tsunami. Acta Psychiatr Scand. 2010 Apr;121(4):289-300. doi: 10.1111/j.1600-0447.2009.01466.x. Epub 2009 Aug 19. PMID 19694633
- [Background] Katzman MA, Vermani M, Gerbarg PL, Brown RP, Iorio C, Davis M, Cameron C, Tsirgielis D. A multicomponent yoga-based, breath intervention program as an adjunctive treatment in patients suffering from generalized anxiety disorder with or without comorbidities. Int J Yoga. 2012 Jan;5(1):57-65. doi: 10.4103/0973-6131.91716. PMID 22346068
- [Background] Doria S, de Vuono A, Sanlorenzo R, Irtelli F, Mencacci C. Anti-anxiety efficacy of Sudarshan Kriya Yoga in general anxiety disorder: A multicomponent, yoga based, breath intervention program for patients suffering from generalized anxiety disorder with or without comorbidities. J Affect Disord. 2015 Sep 15;184:310-7. doi: 10.1016/j.jad.2015.06.011. Epub 2015 Jun 24. PMID 26142611
- [Background] Hamilton-West K, Pellatt-Higgins T, Sharief F. Evaluation of a Sudarshan Kriya Yoga (SKY) based breath intervention for patients with mild-to-moderate depression and anxiety disorders. Prim Health Care Res Dev. 2019 Jun 20;20:e73. doi: 10.1017/S1463423619000045. PMID 32799993
- [Background] Sharma A, Barrett MS, Cucchiara AJ, Gooneratne NS, Thase ME. A Breathing-Based Meditation Intervention for Patients With Major Depressive Disorder Following Inadequate Response to Antidepressants: A Randomized Pilot Study. J Clin Psychiatry. 2017 Jan;78(1):e59-e63. doi: 10.4088/JCP.16m10819. PMID 27898207
- [Background] Seppala EM, Bradley C, Moeller J, Harouni L, Nandamudi D, Brackett MA. Promoting Mental Health and Psychological Thriving in University Students: A Randomized Controlled Trial of Three Well-Being Interventions. Front Psychiatry. 2020 Jul 15;11:590. doi: 10.3389/fpsyt.2020.00590. eCollection 2020. PMID 32760296
- [Background] Goldstein MR, Lewis GF, Newman R, Brown JM, Bobashev G, Kilpatrick L, Seppala EM, Fishbein DH, Meleth S. Improvements in well-being and vagal tone following a yogic breathing-based life skills workshop in young adults: Two open-trial pilot studies. Int J Yoga. 2016 Jan-Jun;9(1):20-6. doi: 10.4103/0973-6131.171718. PMID 26865767
- [Background] Brown RP, Gerbarg PL. Sudarshan Kriya Yogic breathing in the treatment of stress, anxiety, and depression. Part II--clinical applications and guidelines. J Altern Complement Med. 2005 Aug;11(4):711-7. doi: 10.1089/acm.2005.11.711. PMID 16131297
- [Background] Brown RP, Gerbarg PL. Sudarshan Kriya yogic breathing in the treatment of stress, anxiety, and depression: part I-neurophysiologic model. J Altern Complement Med. 2005 Feb;11(1):189-201. doi: 10.1089/acm.2005.11.189. PMID 15750381
- [Background] Seppala EM, Nitschke JB, Tudorascu DL, Hayes A, Goldstein MR, Nguyen DT, Perlman D, Davidson RJ. Breathing-based meditation decreases posttraumatic stress disorder symptoms in U.S. military veterans: a randomized controlled longitudinal study. J Trauma Stress. 2014 Aug;27(4):397-405. doi: 10.1002/jts.21936. PMID 25158633
- [Background] Toschi-Dias E, Tobaldini E, Solbiati M, Costantino G, Sanlorenzo R, Doria S, Irtelli F, Mencacci C, Montano N. Sudarshan Kriya Yoga improves cardiac autonomic control in patients with anxiety-depression disorders. J Affect Disord. 2017 May;214:74-80. doi: 10.1016/j.jad.2017.03.017. Epub 2017 Mar 7. PMID 28285240
- [Background] Janakiramaiah N, Gangadhar BN, Naga Venkatesha Murthy PJ, Harish MG, Subbakrishna DK, Vedamurthachar A. Antidepressant efficacy of Sudarshan Kriya Yoga (SKY) in melancholia: a randomized comparison with electroconvulsive therapy (ECT) and imipramine. J Affect Disord. 2000 Jan-Mar;57(1-3):255-9. doi: 10.1016/s0165-0327(99)00079-8. PMID 10708840
- [Background] Kumar N, Bhatnagar S, Velpandian T, Patnaik S, Menon G, Mehta M, Kashyap K, Singh V, Surajpal. Randomized Controlled Trial in Advance Stage Breast Cancer Patients for the Effectiveness on Stress Marker and Pain through Sudarshan Kriya and Pranayam. Indian J Palliat Care. 2013 Sep;19(3):180-5. doi: 10.4103/0973-1075.121537. PMID 24347909
- [Background] Chandra S, Jaiswal AK, Singh R, Jha D, Mittal AP. Mental Stress: Neurophysiology and Its Regulation by Sudarshan Kriya Yoga. Int J Yoga. 2017 May-Aug;10(2):67-72. doi: 10.4103/0973-6131.205508. PMID 28546676
- [Background] Ghahremani DG, Oh EY, Dean AC, Mouzakis K, Wilson KD, London ED. Effects of the Youth Empowerment Seminar on impulsive behavior in adolescents. J Adolesc Health. 2013 Jul;53(1):139-41. doi: 10.1016/j.jadohealth.2013.02.010. Epub 2013 Apr 16. PMID 23601502
- [Background] Subramanian S, Elango T, Malligarjunan H, Kochupillai V, Dayalan H. Role of sudarshan kriya and pranayam on lipid profile and blood cell parameters during exam stress: A randomized controlled trial. Int J Yoga. 2012 Jan;5(1):21-7. doi: 10.4103/0973-6131.91702. PMID 22346062
- [Background] Kjellgren A, Bood SA, Axelsson K, Norlander T, Saatcioglu F. Wellness through a comprehensive yogic breathing program - a controlled pilot trial. BMC Complement Altern Med. 2007 Dec 19;7:43. doi: 10.1186/1472-6882-7-43. PMID 18093307
- [Background] Korkmaz A, Bernhardsen GP, Cirit B, Koprucu Suzer G, Kayan H, Bicmen H, Tahra M, Suner A, Lehto SM, Sag D, Saatcioglu F. Sudarshan Kriya Yoga Breathing and a Meditation Program for Burnout Among Physicians: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2353978. doi: 10.1001/jamanetworkopen.2023.53978. PMID 38294813
- [Background] West CP, Dyrbye LN, Satele DV, Shanafelt TD. Colleagues Meeting to Promote and Sustain Satisfaction (COMPASS) Groups for Physician Well-Being: A Randomized Clinical Trial. Mayo Clin Proc. 2021 Oct;96(10):2606-2614. doi: 10.1016/j.mayocp.2021.02.028. Epub 2021 Aug 5. PMID 34366134
- [Background] Cheng ST, Tsui PK, Lam JH. Improving mental health in health care practitioners: randomized controlled trial of a gratitude intervention. J Consult Clin Psychol. 2015 Feb;83(1):177-86. doi: 10.1037/a0037895. Epub 2014 Sep 15. PMID 25222798
- [Background] Fendel JC, Burkle JJ, Goritz AS. Mindfulness-Based Interventions to Reduce Burnout and Stress in Physicians: A Systematic Review and Meta-Analysis. Acad Med. 2021 May 1;96(5):751-764. doi: 10.1097/ACM.0000000000003936. PMID 33496433
- [Background] Kiser SB, Sterns JD, Lai PY, Horick NK, Palamara K. Physician Coaching by Professionally Trained Peers for Burnout and Well-Being: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245645. doi: 10.1001/jamanetworkopen.2024.5645. PMID 38607628
- [Background] Hamidi MS, Bohman B, Sandborg C, Smith-Coggins R, de Vries P, Albert MS, Murphy ML, Welle D, Trockel MT. Estimating institutional physician turnover attributable to self-reported burnout and associated financial burden: a case study. BMC Health Serv Res. 2018 Nov 27;18(1):851. doi: 10.1186/s12913-018-3663-z. PMID 30477483
- [Background] Panagioti M, Geraghty K, Johnson J, Zhou A, Panagopoulou E, Chew-Graham C, Peters D, Hodkinson A, Riley R, Esmail A. Association Between Physician Burnout and Patient Safety, Professionalism, and Patient Satisfaction: A Systematic Review and Meta-analysis. JAMA Intern Med. 2018 Oct 1;178(10):1317-1331. doi: 10.1001/jamainternmed.2018.3713. PMID 30193239 (Retraction: PMID 32421149 JAMA Intern Med. 2020 Jul 1;180(7):931)
- [Background] Amutio A, Martinez-Taboada C, Hermosilla D, Delgado LC. Enhancing relaxation states and positive emotions in physicians through a mindfulness training program: A one-year study. Psychol Health Med. 2015;20(6):720-31. doi: 10.1080/13548506.2014.986143. Epub 2014 Dec 8. PMID 25485658
- [Background] West CP, Dyrbye LN, Rabatin JT, Call TG, Davidson JH, Multari A, Romanski SA, Hellyer JM, Sloan JA, Shanafelt TD. Intervention to promote physician well-being, job satisfaction, and professionalism: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):527-33. doi: 10.1001/jamainternmed.2013.14387. PMID 24515493
- [Background] Gootjes L, Franken IH, Van Strien JW. Cognitive emotion regulation in yogic meditative practitioners. J Psychophysiol (2011) 25(2):87-94. 10.1027/0269-8803/a000043
- [Background] Agte VV, Chiplonkar SA. Sudarshan kriya yoga for improving antioxidant status and reducing anxiety in adults. Altern Complement Ther (2008) 14(2):96-100. 10.1089/act.2008.14204
- [Background] Lee, R. M., Draper, M., & Lee, S. (2001). Social connectedness, dysfunctional interpersonal behaviors, and psychological distress: Testing a mediator model. Journal of Counseling Psychology, 48(3), 310-318.
- [Background] Chhatwal J, Fleurence RL. Realizing the Economic Potential of Meditation and Mindfulness Practices in Mental Health Care. Value Health. 2025 Aug;28(8):1141-1144. doi: 10.1016/j.jval.2025.04.2164. Epub 2025 May 6. PMID 40339644